CLINICAL TRIAL: NCT05771662
Title: Multimodal Brain Monitoring as a Prognostic Tool for Intracerebral Hemorrhage - A Prospective Observational Cohort Study.
Brief Title: Multimodal Brain Monitoring as a Prognostic Tool for Intracerebral Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Other Study IDs: ICH-NEUROICU
Record Dates: First submitted 2023-02-08; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To verify if there is an association between advanced multimodal brain monitoring parameters in the first 48h and fist 7 days of admission with intrahospital and six-months functional outcome, even when controlled to other factors that may influence the outcome. Secondary Goals: To describe multimodal neuromonitoring parameters variation in the first seven days of ICH and identify any trends.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous Intracerebral Hemorrhage
* ICU admission in the first 24hours
* Need for intraparenchymal Neuromonitoring
* Over 18 years old

Exclusion Criteria:

* Tumour, Trauma or known Vascular Lesion
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically Ill, Spontaneous Intracerebral Hemorrhage Adult Patients.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Relation between multimodal brain monitoring parameters and outcome. | 6 months
  Association between advanced multimodal brain monitoring parameters of the first 48h of admission and six months functional outcome (Glasgow Outcome Score Extended)

SECONDARY OUTCOMES:
ICH Neuromonitoring Pattern. | 7 days
  Describe multimodal neuromonitoring parameters variation in the first seven days of ICH and identify trends.
ICH Neuromonitoring and Short Term Outcome | 28 days
  Association between advanced multimodal brain monitoring parameters and 28 days functional outcome (Glasgow Outcome Score Extended)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar São João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No